CLINICAL TRIAL: NCT00640679
Title: Prospective, Randomized, Double-Blind Trial of Abrupt and Tapered Interruption of Long-term Clopidogrel Therapy After Implantation of a Drug-Eluting Stent
Brief Title: Abrupt Versus Tapered Interruption of Chronic Clopidogrel Therapy After DES Implantation
Acronym: ISAR-CAUTION
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to slow enrollment the study was stopped prematurely.
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GE IDE No. A01308
Record Dates: First submitted 2008-03-17; First posted 2008-03-21 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Disease
Keywords: Clopidogrel; Drug-eluting Stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clopidogrel Tapering (Active Comparator)
  Interventions: Drug: Clopidogrel Tapering
- Abrupt Clopidogrel Interruption (Active Comparator)
  Interventions: Drug: Abrupt Clopidogrel Interruption

INTERVENTIONS:
Drug: Abrupt Clopidogrel Interruption — Patients assigned to this group will receive Clopidogrel 75mg per day for an additional period of 4 weeks. Afterwards they will stop the drug abruptly.
  Other Names: Plavix
  Arms: Abrupt Clopidogrel Interruption
Drug: Clopidogrel Tapering — Patients assigned to this group will have Clopidogrel gradually decreased according to a fixed tapering schema of Clopidogrel and Placebo over 4 weeks.
  Other Names: Plavix
  Arms: Clopidogrel Tapering

SUMMARY:
The hypothesis to be tested is that gradual clopidogrel therapy cessation is associated with a superior clinical outcome compared with abrupt cessation (superiority hypothesis).

DETAILED DESCRIPTION:
A possible rebound in platelet activity after clopidogrel withdrawal has been suggested in patients on chronic clopidogrel therapy. However, a systematic evaluation of the role of rapid thienopyridine withdrawal on ischemic complications in patients with treated coronary artery disease has not been addressed by specifically designed studies. The objective of this study is to evaluate the safety and efficacy of abrupt or tapered interruption of chronic clopidogrel therapy after intracoronary drug-eluting stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with planned interruption of chronic clopidogrel therapy after DES implantation
* Informed, written consent by the patient

Exclusion Criteria:

* Planned surgery within the next month
* Active bleeding as reason for clopidogrel discontinuation
* Concomitant coumadin therapy
* Pregnancy (present, suspected or planned) or positive pregnancy test (In women with childbearing potential a negative pregnancy test is mandatory)
* Malignancies or other comorbid conditions with a life expectancy of less than one year or that may result in protocol noncompliance.
* Patient's inability to fully comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2008-04; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Composite of cardiac death, myocardial infarction, stent thrombosis, stroke, major bleeding or rehospitalization due to acute coronary syndrome. | 3 months after randomization

SECONDARY OUTCOMES:
The individual components of the primary endpoint. All cause mortality. | 3 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, MD, Study Chair — Deutsches Herzzentrum Muenchen; Julinda Mehilli, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (2):
- Germany (2):
  - Deutsches Herzzentrum Muenchen, Munich
  - Medizinische Klinik, Klinikum rechts der Isar, Munich

REFERENCES:
- [Result] Fiedler KA, Mehilli J, Kufner S, Schlichting A, Ibrahim T, Sibbing D, Ott I, Schunkert H, Laugwitz KL, Kastrati A, Schulz S. Randomised, double-blind trial on the value of tapered discontinuation of clopidogrel maintenance therapy after drug-eluting stent implantation. Intracoronary Stenting and Antithrombotic Regimen: CAUTION in Discontinuing Clopidogrel Therapy--ISAR-CAUTION. Thromb Haemost. 2014 Jun;111(6):1041-9. doi: 10.1160/TH13-11-0900. Epub 2014 Mar 13. PMID 24633406